CLINICAL TRIAL: NCT06421662
Title: The Effect of Attachment Training Given to Pregnant Women on Mother Infant Attachment
Brief Title: The Role of Attachment Training in Mother-infant Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, GÜVEN BEKTEMUR, Assoc.Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: mother-infant attachment
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Mother-Infant Interaction; Infant Development; Maternal Behavior
Keywords: infant; maternal attachment; attachment training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Thirty pregnant women between 28th and 38th gestational weeks who applied to the outpatient clinic of a training and research hospital were included in the study group. During the training, 7 participants were excluded due to premature birth.
  Interventions: Behavioral: Attachment Training
- Control Group (No Intervention): Thirty-one pregnant women between 28th and 38th gestational weeks who applied to the outpatient clinic of a training and research hospital were included in the control group. The control group was administered only the "Maternal Attachment Inventory " developed by Mary Muller in 1994 and the Turkish validity and reliability study was conducted by Şirin and Kavlak at the 8th week after birth.

INTERVENTIONS:
Behavioral: Attachment Training — The study group was trained online by a psychologist on attachment in two sessions. In order to measure the level of attachment knowledge before and after the training, a test form prepared by the researcher based on the literature and expert opinion was used as pre-test and post-test. In the 8th week after delivery, "Maternal Attachment Inventory " developed by Mary Muller in 1994 and Turkish validity and reliability study was conducted by Şirin and Kavlak.
  Arms: Study Group

SUMMARY:
The study aimed to investigate the effect of attachment training given to pregnant women on mother-infant attachment.Primiparous pregnant women between 28.-38. weeks were randomized into two groups. Pregnant women in the study group were given attachment training for 15 days and the effect of the training on mother-infant attachment was investigated by using the mother-infant attachment scale at postpartum week 8 in comparison with the control group.

DETAILED DESCRIPTION:
Pregnant women between 28th and 38th weeks of gestational age who applied to an outpatient clinic of a training and research hospital were randomized into two groups. The study group was trained online by a psychologist on attachment in two sessions. In order to measure the level of attachment knowledge before and after the training, a test form prepared by the researcher based on the literature and expert opinion was applied as pre-test and post-test. In the 8th week after delivery, "Maternal Attachment Inventory" developed by Mary Muller in 1994 and Turkish validity and reliability study was conducted by Şirin and Kavlak. Maternal Attachment Inventory, Each item contains direct expressions and is always scored as follows: (a)= 4 points, frequently (b)= 3 points, sometimes (c)= 2 points, and never (d)= 1 point. A general score is obtained from the sum of all items. A high score indicates a high level of maternal attachment. The total score from the scale ranges from a minimum of 26 to a maximum of 104

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old with a primiparous pregnancy,
* 28 to 38 weeks of gestation,
* At least primary school graduate,
* Who can use the internet actively and can receive planned training online,
* Can speak and understand Turkish like a native speaker,
* Expectant mothers who voluntarily accepted the study.

Exclusion Criteria:

* Transferring the pregnant woman to another hospital for follow-up and treatment
* Those who cannot use active internet and will not be able to receive online education
* Not completing the post-test after the training
* Not completing the postpartum maternal attachment scale
* Expectant mothers receiving psychiatric treatment
* Those with risky pregnancies
* Any congenital anomaly in the baby
* Unwanted baby status
* Withdrawal of the candidate from the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Primiparous pregnant women
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment | 10 minutes
  Maternal Attachment Inventory (MAI) Each item contains direct expressions and is always scored as follows: (a)= 4 points, frequently (b)= 3 points, sometimes (c)= 2 points, and never (d)= 1 point. A general score is obtained from the sum of all items. A high score indicates a high level of maternal attachment. The total score from the scale ranges from a minimum of 26 to a maximum of 104.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No